CLINICAL TRIAL: NCT05495971
Title: Extended Depth of Focus Contact Lenses for Presbyopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visioneering Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VTI-2206
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Presbyopia
Keywords: soft contact lens
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: Subjects will serve as their own control using objective baseline data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Presbyopia (Experimental): Subject's baseline vision will be compared with vision wearing treatment product
  Interventions: Device: NaturalVue Multifocal

INTERVENTIONS:
Device: NaturalVue Multifocal — EDOF

SUMMARY:
VTI has an FDA cleared soft contact lens product. Its optical design creates an enhanced depth of focus (EDOF), which provides clear distance, intermediate, and near vision. This study is to quantify the enhanced depth of focus and visual impact.

DETAILED DESCRIPTION:
This study will develop defocus curves for Baseline best corrected spectacle refraction and then for the EDOF lens used in this study. A comparison of thge depth of focus for each condition will be made.

ELIGIBILITY:
Inclusion Criteria:

* Suitable and able to wear contact lenses
* Normal best corrected vision (20/25 or better)
* Need reading add +2.00 or stronger

Exclusion Criteria:

* Pre-existing ocular condition that would contraindicating lens wear

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas P. Benoit, OD, Study Director — Visioneering Technologies, Inc
Locations (1):
- VTI, Alpharetta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tuan KA, Benoit DP, O'Connor B. Evaluation of the Functional Visual Range of a Catenary Curve-Based, Extended Depth-of-Focus Contact Lens for Presbyopia. Clin Ophthalmol. 2024 Jul 19;18:2113-2123. doi: 10.2147/OPTH.S468699. eCollection 2024. PMID 39055378

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Presbyopia
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Presbyopia
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 59.2 [51 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 24
Visual acuity [Mean (Standard Deviation); unit: logMAR] — logMAR visual acuity
  logMAR | -0.07 (0.07)

OUTCOME MEASURES:

1. Primary Outcome: LogMAR Visual Acuity
Description: High contrast/high illumination distant (6M) logMAR vision
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Presbyopia
Number analyzed (Participants) | 24
logMAR | -0.07 (0.07)

ADVERSE EVENTS:
Time Frame: 4 hours
Description: Regular investigator assessment
Arm/Group | Presbyopia
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT05495971/Prot_SAP_000.pdf